CLINICAL TRIAL: NCT06450665
Title: Reducing Social Avoidance Among Adolescents With Special Educational Needs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHEN Xiaohua Sylvia, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSEARS20240214005
Record Dates: First submitted 2024-06-05; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Social Avoidant Behavior; Social Anxiety
Keywords: Social Avoidant Behavior; Adolescents; Special Education Needs

STUDY DESIGN:
Intervention Model Description: The intervention group will go through three 30-minute VR sessions over a period of 3 weeks. The wait-list control group will complete the questionnaires in the same interval as the intervention group, with promise of receiving VR intervention after 1-month follow-up is over.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Social Avoidance Intervention (Experimental): The intervention group will go through three 30-minute VR sessions over a period of 3 weeks. Participants will need to complete a baseline survey before the VR sessions and a post-intervention survey after the VR sessions, as well as a 1-month follow-up survey.
  Interventions: Behavioral: VR Social Avoidance Intervention
- Waitlist Control (No Intervention): The wait-list control group will complete the questionnaires in the same interval as the intervention group, with promise of receiving VR intervention after 1-month follow-up is over.

INTERVENTIONS:
Behavioral: VR Social Avoidance Intervention — The intervention is based on cognitive-behavioral approach with a virtual coach acting as the therapist. It will be designed in tandem with input from Hong Kong users to ensure the scenario can resonate with them. By testing beliefs that inhibit confidence in a safe and controlled environment, participants will complete tasks with increasing difficulty in three VR scenarios and learn that they can cope in situations that they previously avoid.
  Arms: VR Social Avoidance Intervention

SUMMARY:
The goal of this clinical trial is to examine the effectiveness of a Virtual Reality (VR) social avoidance intervention in reducing social avoidance symptoms among adolescents with special educational needs. Participants will complete tasks in the VR scenario with increasing difficulty and learn that they can cope in situations that they previously avoid. We hypothesize that, comparing with usual care (i.e. waitlist control), the intervention group will experience a significant reduction on social avoidance symptoms after treatment and this benefit will persist till 1-month follow-up.

DETAILED DESCRIPTION:
Over the past 25 years, VR has been used to complement therapist-delivered psychological interventions, primarily exposure therapy for anxiety related disorders. VR renders real-world social interactions simulation, which allows users to experience an anxiety provoking situation with a greater sense of control. In Hong Kong, with the lack of mental health professionals being a perennial problem, VR-based interventions offer the potential to substantially reduce the treatment time and cost, as well as to increase access to evidence-based psychological interventions.

The Virtual Reality (VR) social avoidance intervention used in the current study is designed based on cognitive-behavioral approach with a virtual coach acting as the therapist. It is designed in tandem with input from Hong Kong users to ensure the scenario can resonate with them.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-19
* Can read traditional Chinese and understand Cantonese
* Self-report on experiencing social avoidance symptoms

Exclusion Criteria:

* History of photosensitive epilepsy
* Impairment of stereoscopic vision
* Balance problems

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 208 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 1st week, 4th week, 8th week
  To assess the extent to which respondents are bothered by depression related symptoms using a 4-point Likert scale from 0 (not at all) to 3 (nearly every day), with higher score indicating higher level of depressive symptoms.
Generalized Anxiety Disorder Assessment (GAD-7) | 1st week, 4th week, 8th week
  To assess the extent to which respondents are bothered by anxiety related symptoms using a 4-point Likert scale from 0 (not at all) to 3 (nearly every day), with higher score indicating higher level of anxiety symptoms.
Work and Social Adjustment Scale (WSAS) | 1st week, 4th week, 8th week
  An adapted version of the 5-item WSAS will be used to measure the extent to which respondents' psychological problem impact their various aspects of life. It is rated on an 8-point Likert scale ranges from 0 (not at all impaired) to 8 (severely impaired). Higher score indicates higher level of impact on various aspects of life caused by psychological problems.
Brief Fear of Negative Evaluation Scale (bFNE) | 1st week, 4th week, 8th week
  This is a 12-item scale that measures the fear associated with being evaluated unfavorably while anticipating or participating in a social situation, including apprehension about receiving negative evaluation, avoidance of being evaluated, and the expectation of being negatively evaluated with a 5-point Likert-type rating scale, ranging from 1 (not at all characteristic of me) to 5 (extremely characteristic of me). Higher score indicates higher level of fear of Negative Evaluation.
Oxford Behavioural Avoidance Task - HK (OBAT-HK) | 1st week, 4th week, 8th week
  This is a 16-item scale, a local adaptation of Freeman's OBAT to assess the extent of which participants feel anxious in everyday situations, and the extent to which they try to avoid those situations. Examples of the situations are: approach another pedestrian to ask for direction, ask the bus driver about which stop you should get off, etc. Participants first answer a question concerning if they could do a specific task right now and then rate the level of distress if they have to perform the task straightaway from 0 (no distress) to 10 (extremely distress), with higher score indicating higher level of social anxiety.
Social phobia (SPS-6) | 1st week, 4th week, 8th week
  This 6-item scale (Peters et al., 2012), which is a shortened version of the 20-item SPS (Mattick & Clarke, 1998), measures individuals' self-report anxiety associated with the performance of various tasks while being scrutinized by others (e.g., working, eating, drinking, writing, using public toilets). It runs on a 5-point Likert scale from 0 (not at all characteristics or true of me) to 4 (extremely characteristics or true of me), with higher score indicating higher tendency of social phobia.
Mental health related Quality of Life (REQoL-20) | 1st week, 4th week, 8th week
  The 20-item scale measures quality of life with positively and negatively worded items in seven themes: activity, hope, belonging and relationships, self-perception, well-being, autonomy, and physical health. The item responses were captured on a five-point Likert scale ranging from 0 (none of the time) to 4 (most or all of the time).
Self-esteem (RSE) | 1st week, 4th week, 8th week
  Rosenberg's Self-Esteem Scale is the standard measure of self-esteem in psychological research. It is composed of 10 items, 5 of which are negatively worded. Scale point ranges from 1="strongly agree" to 4="strongly disagree".
Social Interaction Anxiety Scale-6 (SIAS-6) | 1st week, 4th week, 8th week, and after each session of VR intervention
  This 6-item scale (Peters et al., 2012), which is a shortened version of the 20-item SIAS (Mattick, & Clarke, 1998), measures individuals' self-report distress when interacting with others. It runs on a 5-point Likert scale from 0 (not at all characteristics or true of me) to 4 (extremely characteristics or true of me), with higher score indicating higher tendency of social interaction anxiety.
Social Anxiety Session Change Index (SASCI) | After each session of VR intervention
  An adapted version of the 4-item SASCI will be used to track the intermediate changes for the VR sessions (i.e., a per session update of improvement/ deterioration of level of social avoidance) on four dimensions: anxiety, avoidance, concern about humiliation and embarrassment, and interference, using a 7-point Likert-type scale ranging from 1 (much less than the start of treatment) to 4 (not different from the start of treatment) to 7 (much more than the start of treatment), with lower score indicating less anxiety after the treatment.
Working Alliance Inventory applied to VR and AR (WAI-VAR) | 4th week
  This is a 12-item scale designed to assess therapeutic alliance between the virtual/augmented reality program and the users. Scale points range from 1 (never) to 7 (always), with higher score indicating higher level of adaptation to the VR environment.
Gatineau Presence Questionnaire (GPQ) | 4th week
  This is a 4-item scale (Laforest et al., 2016) designed to assess the feeling of presence experienced in a virtual environment. Sample items include "the impression of being here", "appraising the experience as being real". Scale point ranges from 0 to 100, with higher score indicating more feeling of presence experienced in a virtual environment.
Social presence (SPSQ) | 4th week
  The five-item social presence questionnaire measures how much participants perceived the virtual human in the room to be like an actual person. Participants rated on a Likert-type scale (from -3 to +3). A positive social presence score indicates that the participant perceived the virtual human as conscious and aware, whereas a negative score indicates that the participant perceived the virtual human as unconscious and unaware.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Sylvia Chen, Principal Investigator — The Hong Kong Polytechnic University; Winnie Wing Sze Mak, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Applied Social Sciences, PolyU, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Topper, M., Emmelkamp, P. M., & Ehring, T. (2010). Improving prevention of depression and anxiety disorders: Repetitive negative thinking as a promising target. Applied and Preventive Psychology, 14, 57-71.
- [Background] Choi EPH, Hui BPH, Wan EYF. Depression and Anxiety in Hong Kong during COVID-19. Int J Environ Res Public Health. 2020 May 25;17(10):3740. doi: 10.3390/ijerph17103740. PMID 32466251
- [Background] Freeman D, Haselton P, Freeman J, Spanlang B, Kishore S, Albery E, Denne M, Brown P, Slater M, Nickless A. Automated psychological therapy using immersive virtual reality for treatment of fear of heights: a single-blind, parallel-group, randomised controlled trial. Lancet Psychiatry. 2018 Aug;5(8):625-632. doi: 10.1016/S2215-0366(18)30226-8. Epub 2018 Jul 11. PMID 30007519
- [Background] Riva G. Virtual reality in psychotherapy: review. Cyberpsychol Behav. 2005 Jun;8(3):220-30; discussion 231-40. doi: 10.1089/cpb.2005.8.220. PMID 15971972
- [Background] Martingano, A. J., Hererra, F., & Konrath, S. (2021). Virtual reality improves emotional but not cognitive empathy: A meta-analysis. Technology, Mind, and Behavior. http://doi.org/10.1037/tmb0000034
- [Background] Van Kerrebroeck, H., Brengman, M., & Willems, K. (2017). When brands come to life: experimental research on the vividness effect of Virtual Reality in transformational marketing communications. Virtual Reality, 21(4), 177-191. http://doi.org/10.1007/s10055-017-0306-3
- [Result] Peters L, Sunderland M, Andrews G, Rapee RM, Mattick RP. Development of a short form Social Interaction Anxiety (SIAS) and Social Phobia Scale (SPS) using nonparametric item response theory: the SIAS-6 and the SPS-6. Psychol Assess. 2012 Mar;24(1):66-76. doi: 10.1037/a0024544. Epub 2011 Jul 11. PMID 21744971
- [Result] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Result] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Result] Keetharuth AD, Brazier J, Connell J, Bjorner JB, Carlton J, Taylor Buck E, Ricketts T, McKendrick K, Browne J, Croudace T, Barkham M. Recovering Quality of Life (ReQoL): a new generic self-reported outcome measure for use with people experiencing mental health difficulties. Br J Psychiatry. 2018 Jan;212(1):42-49. doi: 10.1192/bjp.2017.10. PMID 29433611
- [Result] Weeks JW, Heimberg RG, Fresco DM, Hart TA, Turk CL, Schneier FR, Liebowitz MR. Empirical validation and psychometric evaluation of the Brief Fear of Negative Evaluation Scale in patients with social anxiety disorder. Psychol Assess. 2005 Jun;17(2):179-90. doi: 10.1037/1040-3590.17.2.179. PMID 16029105
- [Result] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Result] Freeman, D., & Lambe, L. (2019b). Self-Report: Oxford Behavioural Avoidance Task, version 2. University of Oxford.
- [Result] Rosenberg, M. (1965). Rosenberg self-esteem scale (RSE). Acceptance and Commitment Therapy. Measures Package, 61.
- [Result] Miragall M, Banos RM, Cebolla A, Botella C. Working alliance inventory applied to virtual and augmented reality (WAI-VAR): psychometrics and therapeutic outcomes. Front Psychol. 2015 Oct 8;6:1531. doi: 10.3389/fpsyg.2015.01531. eCollection 2015. PMID 26500589
- [Result] Laforest, M., Bouchard, S., Crétu, A., & Mesly, O. (2016). Inducing an Anxiety Response Using a Contaminated Virtual Environment: Validation of a Therapeutic Tool for Obsessive-Compulsive Disorder. Frontiers In ICT, 3. https://doi.org/10.3389/fict.2016.00018
- [Result] Bailenson JN, Blascovich J, Beall AC, Loomis JM. Interpersonal distance in immersive virtual environments. Pers Soc Psychol Bull. 2003 Jul;29(7):819-33. doi: 10.1177/0146167203029007002. PMID 15018671
- [Result] Hayes SA, Miller NA, Hope DA, Heimberg RG, Juster HR. Assessing Client Progress Session by Session in the Treatment of Social Anxiety Disorder: The Social Anxiety Session Change Index. Cogn Behav Pract. 2008 May 1;15(2):203-2011. doi: 10.1016/j.cbpra.2007.02.010. PMID 25075171